CLINICAL TRIAL: NCT05992610
Title: Induction Treatment in Patients With Squamous Cell Carcinoma (SCC) of the Head and Neck Region Consisting Concomitant Chemotherapy and Low-dose Ionizing Radiotherapy
Brief Title: Induction Treatment in SCC of the Head and Neck Region - Concomitant Chemotherapy and Low-dose Radiotherapy
Acronym: iCHRTL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: iCHRTL
Record Dates: First submitted 2023-03-13; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-03

CONDITIONS: Squamous Cell Carcinoma of Oral Cavity; Pharynx Carcinoma; Larynx Carcinoma; Paranasal Sinus Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Pharyngeal Neoplasms; Laryngeal Neoplasms; Paranasal Sinus Neoplasms | interventions — Drug Therapy; CP protocol

STUDY DESIGN:
Intervention Model Description: Interventional, open, allocation to concomitant chemotherapy and low-dose ionizing radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy (Ch)+ Radiotherapy (RT) (Experimental): Induction phase:
  Chemotherapy based on carboplatin 6 AUC (area under the curve) + paclitaxel 75 mg/m2 carboplatin 6 AUC 30-minute infusion on D: 1 (maximum carboplatin dose is 700 mg) paclitaxel 75 mg/m2 1-hour infusion on D: 1, 8, 15
  Radiotherapy:
  D:1 - 2 x 0,5 Gy (first dose up to one hour after the end of the carboplatin infusion, second dose 3 to 6 hours later), D:2 - 2 x 0,5 Gy (interval between doses not less than 3 hours), D:8 and D:15 - 2 x 0,5 Gy (first dose up to one hour after the end of the chemotherapeutic infusion, second dose 3 to 6 hours later).
  Interventions: Other: Chemotherapy (carboplatin+paclitaxel) with concomitant low dose ionizing radiotherapy

INTERVENTIONS:
Other: Chemotherapy (carboplatin+paclitaxel) with concomitant low dose ionizing radiotherapy — Chemotherapy based on carboplatin 6 AUC + paclitaxel 75 mg/m2.
  Radiotherapy:
  D:1 - 2 x 0,5 Gy (first dose up to one hour after the end of the carboplatin infusion, second dose 3 to 6 hours later), D:2 - 2 x 0,5 Gy (interval between doses not less than 3 hours), D:8 and D:15 - 2 x 0,5 Gy (first dose up to one hour after the end of the chemotherapeutic infusion, second dose 3 to 6 hours later).

SUMMARY:
Non-commercial clinical study to assess:

1. efficacy of iCHRTL in patients with advanced squamous cell carcinoma of oral cavity, pharynx carcinoma, larynx carcinoma or paranasal sinus carcinoma.
2. tolerability of iCHRTL in patients with advanced squamous cell carcinoma of oral cavity, pharynx carcinoma, larynx carcinoma or paranasal sinus carcinoma.
3. molecular and biochemical effect of low doses of ionizing radiation.

DETAILED DESCRIPTION:
40 patients with squamous cell carcinoma of oral cavity, pharynx, larynx or paranasal sinuses in stage III or IV, previously not treated for this reason and eligible for induction chemotherapy.

Study treatment:

Induction phase:

Chemotherapy based on carboplatin 6 area under the curve (AUC) + paclitaxel 75 mg/m2 carboplatin 6 AUC 30-minute infusion on D: 1 (maximum carboplatin dose is 700 mg) paclitaxel 75 mg/m2 1-hour infusion on D: 1, 8, 15

Radiotherapy:

D:1 - 2 x 0,5 Gy (first dose up to one hour after the end of the carboplatin infusion, second dose 3 to 6 hours later), D:2 - 2 x 0,5 Gy (interval between doses not less than 3 hours), D:8 and D:15 - 2 x 0,5 Gy (first dose up to one hour after the end of the chemotherapeutic infusion, second dose 3 to 6 hours later).

2 cycles of induction treatment are planned. Interval between the last day of cycle I and the first day of cycle II is 7 days. After 2 weeks from second cycle Positron emission tomography (PET) and Magnetic Resonance (MR), medical case conference and qualification to further treatment: Radiotherapy (RT), Chemo-radiotherapy (CHRT) or other, depending on the medical decision.

Planned based on the optimal technique for a particular clinical case preferred: Intensity Modulated Radiation Therapy (IMRT). Preparation of IMRT plan will be based on computed tomography (CT) scans. Early tolerance of radiotherapy will be assessed for local reaction. At least once every 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with squamous cell carcinoma of oral cavity, upper, middle, lower pharynx carcinoma, larynx carcinoma or paranasal sinus carcinoma in advanced stage III or IV and previously not treated for this reason.
2. Severity of the disease: N1 > 2 cm, N2, N3 ; T2, T3, T4, M0
3. Patient eligible for radical treatment with induction chemotherapy (at least in good general condition (ZUBROD 0-1) with no significant additional diseases disqualifying from induction chemotherapy).
4. Written informed consent form to the proposed therapeutic scheme.
5. Age over 18 years.

Exclusion Criteria:

1. Subjects with known or suspected hypersensitivity to any of the study mediations.
2. Baseline values for the following parameters (in the screening phase):

   * Creatinine >2,0 x upper limit of normal (ULN) - unless creatinine clearance is normal
   * Total bilirubin >1,5 x ULN (except for hyperbilirubinemia caused by Gilbert's syndrome)
   * Alanine Transaminase (ALT) activity, Aspartate Transaminase (ASPAT) >2,5 x ULN
   * Alkaline phosphatase activity >2,5 x ULN
3. Prior treatment with any unauthorized medication or investigational treatment before the 5 half-lives of that substance or 4 weeks prior to study entry (a longer period of time should be assumed), or subjects currently enrolled to other interventional clinical trials.
4. Concomitant malignancy or history of a malignancy with a significant potential impact to tolerability or effectivity of iCHRTL.
5. Chronic or active infection requiring antibiotic, antifungal or antiviral treatment, such as, but not limited to: chronic kidney infection, chronic respiratory tract infection with bronchospasm, tuberculosis or active hepatitis C virus infection.
6. History of significant cerebrovascular disease within 6 months or currently symptomatic or its implications.
7. Human Immunodeficiency Virus (HIV) infection.
8. Clinically significant heart disease including unstable angina, myocardial infarction within 6 months prior to study entry, severe congestive circulatory failure class New York Heart Association (NYHA) III-IV, arrhythmias unless it is treated, except for collateral contractions or minimal conduction disorders.
9. Significant concomitant disease that cannot be treated, such as, but not limited to kidney, liver, gastrointestinal, endocrine system, respiratory, neurological and brain diseases and mental illnesses that may pose a risk to the patient in the opinion of the investigator.
10. Active hepatitis B virus (HBV) infection, defined as having a positive Hepatitis B surface antigen (HBsAg) test. Moreover, in case of a negative HBsAg test result but a positive Hepatitis B core Antibody (HBcAb) test result (regardless of HBsAb status), HBV DNA should be determined and in case of a positive result the patient cannot be included to the study.
11. Active hepatitis C virus (HCV) infection, defined as having a positive Hepatitis C Antibody (HCAb) test, in which case Hepatitis C virus recombinant immunoblot assay (HCV RIBA) should be determined from the same sample to confirm the result.
12. Pregnancy or breastfeeding (women of childbearing potential must have pregnancy test performed during screening).
13. Women of childbearing potential, including women whose last menstrual period occurred in less than one year before screening, who cannot or do not want to use adequate contraception methods from the beginning of the study until 6 months after the last dose of study drug. Adequate contraception is defines as the use of oral hormonal contraceptives, an intrauterine device, a double barrier method or sexual abstinence.
14. Men who cannot or do not want to use adequate contraception methods from the beginning of the study until 6 months after the last dose of study medication.
15. Patients who cannot or do not want to adhere to the study Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) after induction | 1 year post-induction
  Complete+partial response in percent
Objective response rate (ORR) after induction | 3 years post-induction
  Complete+partial response in percent
Loco-regional control (LRC) rate | 1 year post-induction
  Rate of local lesions complete response (CR) +partial response (PR)+stable disease (SD)
Loco-regional control (LRC) rate | 3 years post-induction
  Rate of local lesions CR+PR+SD
Distant metastasis rate | 1 year post-induction
  Rate of patients with distant metastases
Distant metastasis rate | 3 years post-induction
  Rate of patients with distant metastases
Overall survival time (OS) | Date of treatment start - to 1 year
  Rate of death within time from treatment start to 1 year
Overall survival time (OS) | Date of treatment start - to 3 years
  Rate of death within time from treatment start to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Składowski, MD PhD, Study Chair — Maria Sklodowska-Curie National Research Institute of Oncology (MSCNRIO)
Locations (1):
- The Maria Sklodowska-Curie National Research Institute of Oncology, Branch in Gliwice, Gliwice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No